CLINICAL TRIAL: NCT05944523
Title: Comparison of the Effect of Preemptive and Post-operative Erector Spina Plane Block on Intraoperative Opioid Consumption and Postoperative Analgesia in Patients Who Will Undergo Elective Thoracotomy Surgery, Guided by the Nociception Level Index (NoL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Canan Tokur, Research Assistant, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CananT
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Erector Spina Plan Block; Preemptive Analgesia; Thoracotomy; Nociception Level Index(NoL)
Keywords: preemptive analgesia; erector spina plan block; nociception level (NoL) index; thoracotomy; opioid consumption
MeSH Terms: conditions — Erythema Multiforme

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): The group in which preemptive erector spina plane block was applied
  Interventions: Procedure: Erector Spina Plan Block
- Group 2 (Active Comparator): The group in which the end of the surgery was applied to the erector spina plane block
  Interventions: Procedure: Erector Spina Plan Block

INTERVENTIONS:
Procedure: Erector Spina Plan Block — Preemptive erector spina plan block and postoperative erector spina plan block were applied to patients undergoing thoracotomy. The effect of the time of application on intraoperative opioid consumption was compared with the Nociception Level Index pain monitor.

SUMMARY:
The patients who will participate in the study will be determined and informed according to the inclusion and exclusion criteria, and the patients who signed the informed consent form will be included in the study.52 patients who will undergo elective thoracotomy surgery will be divided into double-blinded 2 sided as preemptive and postoperative erector spina plane block.

Intraoperative pain status of the patients will be determined by the "Nociception Level Index" device and analgesia will be provided with fentanyl. The primary aim of the study is to compare the intraoperative opioid consumption of two groups with plan block at different times.

In the postoperative period, patient-controlled analgesia device will be given to both groups for rescue analgesia. The opioid consumption of the patients will be controlled in this way in the postoperative period and their pain status will be determined. The secondary aim of the study is to examine the effect of plan block application time on the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* ASA classification <4
* No history of allergy or hypersensitivity to the drugs we use throughout the procedure
* BMI ≤ 35
* No history of neuropathy
* Surgeries other than emergency surgery
* Volunteer for the study
* No presence of infection at the injection site
* No any pyschiatric disease that would prevent the evaluation of the pain score

Exclusion Criteria:

* Under the age of 18 or over the age of 65
* ASA classification ≥ 4
* History of allergy or hypersensitivity to the drugs we use throughout the procedure
* BMI > 35
* History of neuropathy
* Undergoing emergency surgery
* Not be a volunteer for the study
* Presence of infection at the injection site
* Having a pyschiatric disease that would prevent the evaluation of the pain score
* Pregnancy
* Undergo surgery again during the postoperative follow-up period for any reason

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The value of Nociception Level Index (NoL) in both preemptive and postoperative groups | Up to 24 hours
  We aim to determine the effect of preemptive or postoperative application of ESPB ın the amount of intraopioid consumption by Nociception Level Index

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Alkış, Prof. Dr., Study Director — Faculty of Medicine, Ankara University
Locations (1):
- Faculty of Medicine, Ankara University, Ankara, Turkey (Türkiye)